CLINICAL TRIAL: NCT00488566
Title: Double Blind, Randomised, Placebo Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Doses of GSK Drug and the Effect of Single Doses of GSK Drug or Lamotrigine on Resting Motor Threshold in Healthy Volunteers
Brief Title: GSK Drug Single Dose Escalation And Their Effect On Resting Motor Threshold In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SCB107718
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder,; single doses,; resting motor threshold; TMS,
MeSH Terms: conditions — Bipolar Disorder | interventions — vixotrigine; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Other): Single dose escalation
  Interventions: Drug: GSK drug; Other: Placebo
- Part 2 (Other): Pharmacodynamic assessment
  Interventions: Drug: GSK drug; Other: Placebo; Other: Lamictal

INTERVENTIONS:
Drug: GSK drug — GSK drug
  Other Names: BIIB074 and CNV1014802
Other: Placebo — Placebo
Other: Lamictal — Positive control
  Arms: Part 2

SUMMARY:
This is a First Time in Human Study to assess the safety, tolerability, pharmacokinetics and resting motor threshold (rMT) of single doses of GSK drug in healthy volunteers.This will be a 2 part and 2 centre study.Part 1 will be a double-blind, randomized, placebo-controlled, single oral dose, dose-rising, cross-over study in healthy male and female (of non-child bearing potential) volunteers.Subjects will be randomized into cohorts of 10 subjects and cohorts will be recruited until the pre-defined safety or PK stopping limits are reached.Each subject will receive placebo and no more than 4 ascending doses of GSK drug in a randomized sequence on 5 separate study occasions.Each dosing session will take place over 2 days and there will be at least one subject on placebo on each day. There will be only one subject on any new active dose during the first day.Part 2 will be a randomised, double-blind, double-dummy, placebo-controlled, cross-over study to investigate the effect of single doses of GSK drug and lamotrigine on resting motor threshold in healthy male subjects. Subjects will attend the unit a maximum of 4 separate occasions.During each session subjects will receive up to 4 TMS measurements and single doses of either GSK drug, lamotrigine or placebo, in a randomised manner.Up to two doses of GSK drug will be investigated.

DETAILED DESCRIPTION:
This study, previously posted by GlaxoSmithKline (GSK), was transitioned to Convergence Pharmaceuticals, Ltd., which spun off from GSK. Convergence Pharmaceuticals, Ltd., has now been acquired by Biogen.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* Healthy male subjects aged between 18 and 65 yrs and female (of non-child bearing potential) subjects aged between 18 and 50 years.

Part 2 Inclusion Criteria:

* right-handed healthy male subjects aged between 18 and 65 years.

Parts 1 & 2 Inclusion Criteria:

* body weight >50 kg and Body Mass Index (BMI) within the range 19 - 29.9 kg/m2 inclusive.
* No abnormality on relevant clinical examination.
* No abnormality on relevant clinical chemistry or haematology examination at the pre-study medical examination.
* A 12-lead ECG at the pre-study medical examination which is normal.
* Non-smokers.
* Signed and dated written informed consent prior to any study procedures being done.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Parts 1&2 Exclusion Criteria:

* exceeding weekly recommended alcohol intake.
* An unwillingness of a male subject to use a condom/ spermicide in addition to having their female partner use another form of contraception.
* A positive Hepatitis B surface antigen, Hepatitis C antibody, and Human Immunodeficiency Virus (HIV) antibody result at screening.
* A positive urine drug test at screening or prior to each treatment period.
* History of alcohol/drug abuse or dependence within 12 months of the study.
* Urine cotinine levels indicative of smoking.
* History or regular use of tobacco or nicotine containing products within 6 months prior to screening.
* QTc interval > 450 ms.
* Current or past history of symptomatic orthostatic hypotension. Sitting systolic blood pressure >139 or <90 mmHg and/or diastolic blood pressure >100 or <50 mmHg. Standing heart rate <45 bpm.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dose of current study medication. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of moderate/high tyramine containing food or drinks from 1 week prior to the first dose and until discharge, following the last dose.
* History of hypersensitivity to lamotrigine.
* History of sensitivity to any of the study medications, or components thereof.Or a history of drug, cosmetic or other allergy that, in the opinion of the physician, might interfere with the conduct of the study.
* History of known or suspected seizures, including infantile febrile, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits).
* Where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.

Part 2 Exclusion Criteria:

* History of clinically relevant skin rashes and allergies.
* Poorly-controlled migraine headaches.
* Implanted metal devices including pacemakers.
* Previous brain neurosurgery.
* History of neurological disorders and stroke.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-05-31 (Actual); Primary Completion 2008-05-31 (Actual); Study Completion 2008-05-31 (Actual)

PRIMARY OUTCOMES:
Part1:AEs for the duration of the study; | duration of the study
ECG,vitals and MAO activity predose and upto 48h post dose; | predose and upto 48h post dose
clinical labs predose and upto 24h post dose. | predose and upto 24h post dose
PK parameters up to 48h post dose. | up to 48h post dose
Part2:Difference in rMT between pre-and post-dose and relationship with PK. | between pre-and post-dose and relationship with PK

SECONDARY OUTCOMES:
Part1:Bond-Lader and body sway predose and upto 24h postdose. | predose and upto 24h postdose
Part2:AEs for the duration of the study;. | duration of the study
ECG,vitals and MAO activity predose and upto 48h postdose; | predose and upto 48h postdose
clinical labs predose and upto 24h postdose | predose and upto 24h postdose

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Medical Director, Study Director — Biogen
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, London